CLINICAL TRIAL: NCT04177199
Title: Prospective Triage HF+ Evaluation: What is the Workload Burden Associated With Using the Triage HF+ Care Pathway?
Brief Title: What is the Workload Burden Associated With Using the Triage HF+ Care Pathway?
Acronym: TRIAGE-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Medtronic (Industry); Pennine Acute Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B00454
Record Dates: First submitted 2019-09-05; First posted 2019-11-26 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: TRIAGE HF Pathway — A new care pathway (Triage-HF Plus) for the remote monitoring and management of heart failure stability in a cohort of device patients at 3 hospital sites in North West England.

SUMMARY:
This observational, prospective real-world evaluation will estimate and characterize the heart-failure related clinical workload burden associated with implementing a new care pathway (Triage-HF Plus) for remote monitoring and management in a cohort of device patients at 3 hospital sites in North West England as compared to the heart-failure related clinical workload burden prior to using this new care pathway. Triage-HF Plus incorporates the Triage-HF algorithm which is a device-based algorithm that uses the input from the integrated device diagnostics to detect changes in physiological parameters which may indicate an individual's increased risk of heart failure event in the 30 days after a high Triage-HF score.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with a Medtronic ICD, CRT-D, or CRT-P device that is Triage-HF compatible and capable of automated transmission. Note: Remote monitoring data will not be available for 60 days post a new or replacement implant but patients can be enrolled in the evaluation any time after implant.
* Patient (or patient's legally authorized representative) is willing and able to provide written informed consent.
* Patients with CareAlerts already turned ON will be included in the prospective part of the evaluation but their data may be excluded from the pre-Triage-HF Plus (current state) data analysis.
* Patients willing and able to have CareLink monitor active at all times.

Exclusion Criteria:

* Patient is enrolled in another conflicting evaluation/study that could confound the results of this evaluation by increasing clinic workload burden for that patient and/or impact clinical interventions and patient outcomes
* All patients with non-Triage-HF compatible devices
* All patients with devices that require manual transmission (non-automated)
* Patient is unwilling or unable to comply with the protocol, including follow-up visits and CareLink transmissions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged > 18 years with Medtronic CareLink® and Triage-HF compatible cardiac device in situ undergoing remote monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of clinical touchpoints will be used to calculate clinical workload burden | Duration of study, expected 18 months
  The workload burden associated with using the Triage HF+ care pathway as compared to the heart failure-related clinic burden prior to using the Triage HF+ care pathway will be calculated using clinical touchpoints including number of hospitalisations, number of A&E/ MAU visits, number of outpatient appointments, number of remote scheduled device follow ups, and number of telephone contacts.
Time for completing clinical touchpoints will be used to calculate clinical workload burden | Duration of study, expected 18 months
  Estimated time for completing clinical touchpoint activities will be calculated from established NHS guidelines/ standards and used to calculate clinical workload burden.

SECONDARY OUTCOMES:
Number of clinical touchpoints pre-Triage-HF Plus (current state) compared to post-Triage-HF Plus Implementation (future state, prospective). | Duration of study, expected 18 months
  Secondary, ancillary metrics (descriptive statistics) will be collected to characterize the clinical context pre-Triage-HF Plus (current state) and post-Triage-HF Plus Implementation (future state, prospective) and guide further improvements. Metrics include total number of Triage HF transmissions, total scheduled transmissions, number of low/ medium/high Triage HF risk scores, number of high Triage HF episodes, number of patients with high Triage HF risk scores, and number of hospitalisations.
Cost of Triage-HF Plus pathway at each site | Duration of study, expected 18 months
  Estimated time for completing clinical touchpoint activities will be calculated from established NHS guidelines/ standards and used to calculate the cost of the Triage HF pathway at each site.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Pennine Acute Hospitals NHS Foundation Trust, Royal Oldham Hospital, Oldham, Lancashire
  - Manchester Royal Infirmary, Manchester University NHS Foundation Trust, Manchester
  - Wythenshawe Hospital, Manchester University NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Ahmed FZ, Harwood R, Lanctin D, Leonard C, Medland S, Afonso D, Mealing S, Weldon T, Blunt C, Campbell NG, Taylor JK. Economic evaluation of the TriageHF Plus clinical pathway for device-based remote monitoring in heart failure. Heart. 2025 Dec 17:heartjnl-2025-326702. doi: 10.1136/heartjnl-2025-326702. Online ahead of print. PMID 41407535
- [Derived] Taylor JK, Ndiaye H, Daniels M, Ahmed F; Triage-HF Plus investigators. Lockdown, slow down: impact of the COVID-19 pandemic on physical activity-an observational study. Open Heart. 2021 Jun;8(1):e001600. doi: 10.1136/openhrt-2021-001600. PMID 34088789